CLINICAL TRIAL: NCT01451450
Title: A Phase II, Randomized, Double Blind, Placebo-controlled, Parallel Design, Dose Ranging, Multi-center Trial of Four Levels of Exposure of QGE031 s.c. for 16 Weeks in Subjects Aged 18-50 Years of Age With Peanut Allergy
Brief Title: Efficacy and Safety of 4 Doses of QGE031 in Patients 18-50 Years of Age With Peanut Allergy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQGE031A2208; 2011-000631-92 (EudraCT Number)
Record Dates: First submitted 2011-10-10; First posted 2011-10-13 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Peanut Allergy
Keywords: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- QGE031 A (Experimental)
  Interventions: Drug: QGE031
- QGE031 B (Experimental)
  Interventions: Drug: QGE031
- QGE031 C (Experimental)
  Interventions: Drug: QGE031
- QGE031 D (Experimental)
  Interventions: Drug: QGE031
- Placebo A (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo B (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo C (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGE031 — QGE031 liquid for subcutaneous injection.
  Arms: QGE031 A; QGE031 B; QGE031 C; QGE031 D
Drug: Placebo — Placebo liquid for subcutaneous injection.
  Arms: Placebo A; Placebo B; Placebo C; Placebo D

SUMMARY:
This study will assess the clinical potency of several exposure levels of QGE031 in decreasing the sensitivity against peanut allergen.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of acute peanut allergy as manifested by urticaria, angioedema, gastro-intestinal or respiratory tract symptoms, with acute onset of symptoms after ingestion (up to 2 hours).
* Positive peanut food challenge at baseline, i.e., have objective allergic events at a level of 300mg (not cumulative) or below of peanut protein but not to the placebo test.

Main Exclusion Criteria:

* Prior exposure to any monoclonal antibody treatment
* Asthma patients on maintenance long acting beta-agonists
* Use of systemic corticosteroids
* Concomitant use of beta blockers, ACE inhibitors, tiotropium or ipratropium, antidepressants, oral beta-agonists
* Use of immunosuppressants within 6 months of visit 1 Other protocol-defined inclusion/exclusion criteria may appy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals